CLINICAL TRIAL: NCT01520181
Title: Extended Open Challenge in Patients With a History of Drug Eruption Following Beta-lactam Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Arnon Goldberg, Head, Allergy and Clinical Immunology Unit, Meir Hospital, Kfar-Saba, Israel, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PEN5
Record Dates: First submitted 2011-11-20; First posted 2012-01-27 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Beta-lactam Allergy

INTERVENTIONS:
Drug: Beta-lactam oral challenge — Oral daily dose, according to patient's weight, of amoxicillin or other suspected beta-lactam will be administered for 5 consecutive days

SUMMARY:
Beta-lactam allergy is the most prevalent drug allergy. Drug eruption is the most common symptom whereas life-threatening anaphylaxis is rather rare. A recently published study (Journal of Allergy and Clinical Immunology, January 2011, Vol. 127, p. 218-222) described the safety of a 2-day oral beta-lactam challenge in penicillin-allergic patients, disregarding their penicillin skin test results. In the proposed study the investigators will similarly challenge beta-lactam allergic patients, both children and adults for an extended (5 days) period of time. The study will include patients with a history of a skin rash following beta-lactam administration as well as patients who cannot provide any data on their presumed allergic reaction, disregarding their penicillin skin test results.

ELIGIBILITY:
Inclusion Criteria:

* History of skin rash following the administration of beta-lactam antibiotic
* Patients with a diagnosis of penicillin allergy who have no data on the nature of the symptoms that have eventually resulted in establishing this diagnosis

Exclusion Criteria:

* Patients in whom the rash appeared within 1 hour after the last dose of the drug
* Patients who also developed other anaphylactic symptoms
* Patients who had a life-threatening rash such as Stevens-Johnson Syndrome, Toxic Epidermal Necrolysis or DRESS.
* Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The safety of a 5-day oral challenge in patients with suspected beta-lactam allergy | 5 days
  In case of the development of any adverse reactions throughout the 5-day challenge patients will notify the investigators over the phone. If assessed necessary by the investigators, patients will return to the Allergy Clinic for repeated evaluation. After completion of the 5-day challenge all patients will be contacted by the investigators and will be inquired about any adverse reactions throughout the challenge. The number of participants with adverse reactions to the challenge will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Arnon Goldberg, Allergy and Clinical Unit, Meir Medical Center, Kfar Saba, Israel